CLINICAL TRIAL: NCT04395183
Title: 31P-MRS and Resting State Functional Connectivity Analysis of the Effects of 5-hydroxytryptophan and Creatine for Antidepressant Augmentation in Patients With SSRI/SNRI-resistant Major Depressive Disorder
Brief Title: 5-HTP and Creatine for Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Brent Michael Kious, MD, PhD, Assistant Professor of Psychiatry, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB_00132830
Record Dates: First submitted 2020-05-15; First posted 2020-05-20 (Actual); Results first posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — 5-Hydroxytryptophan; Creatine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Randomized, double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 5-HTP + Placebo (Active Comparator): 5-hydroxytryptophan 100mg PO BID plus placebo matched to creatine monohydrate
  Interventions: Drug: 5-Hydroxytryptophan 100 MG; Drug: placebo matched to 5-HTP
- Creatine + Placebo (Active Comparator): Creatine 5g PO qday plus placebo matched to 5-HTP
  Interventions: Drug: Creatine monohydrate; Drug: placebo matched to 5-HTP
- Creatine + 5-HTP (Active Comparator): Creatine 5g PO qday plus 5-hydroxytryptophan 100mg PO BID
  Interventions: Drug: 5-Hydroxytryptophan 100 MG; Drug: Creatine monohydrate
- Double Placebo (Placebo Comparator): Creatine-matched placebo and 5-HTP-matched placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 5-Hydroxytryptophan 100 MG — 5-HTP 100mg PO BID
  Other Names: creatine monohydrate
  Arms: 5-HTP + Placebo; Creatine + 5-HTP
Drug: Creatine monohydrate — Creatine monohydrate 5g PO qday
  Arms: Creatine + 5-HTP; Creatine + Placebo
Drug: placebo matched to 5-HTP — placebo matched to 5-HTP
  Arms: 5-HTP + Placebo; Creatine + Placebo
Drug: Placebo — Dextrose either as loose powder (matched to creatine) or encapsulated (matched to 5-HTP)
  Arms: Double Placebo

SUMMARY:
This is a three-armed clinical trial examining the effect of 5-hydroxytryptophan and creatine monohydrate as augmenting agents for the treatment of depression. Subjects will be randomized between 5-HTP + placebo, creatine + placebo, and 5-HTP + creatine, for 8 weeks. The ability of the interventions to affect biomarkers associated with depression will be assessed using brain phosphorus magnetic resonance spectroscopy, functional connectivity imaging, and plasma serotonin levels.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) has a lifetime prevalence of over 16%1 and is associated with reduced work productivity,2 disability,3 increased mortality,4 and increased rates of suicide attempts5 and completed suicides.6 Unfortunately, ~34% fail to respond to standard ADs (ADs).7 Environmental and patient-level factors that increase the risk of MDD could pinpoint novel mechanisms underlying the disorder. One such factor may be relative hypoxia. Persons with hypoxic medical conditions, such as asthma and chronic obstructive pulmonary disease, are at higher risk of depression and suicide compared to those with other chronic medical conditions.8-12 Smoking also promotes hypoxia13 and is linked to increased risks of suicide and depression.14-16 Of special relevance to this study, living at high altitude produces relative hypoxia even after months,17 and is linked to increased risks of suicide18-22 and depression.23,24 Hypoxia could contribute to MDD in at least two ways. First, brain bioenergetics are altered in both hypoxia and MDD. Hypoxia reduces several neurochemical markers of brain activity, including phosphocreatine (PCr) and n-acetylaspartate (NAA),25 and alters mitochondrial dynamics in the hippocampus.26,27 Proton magnetic resonance spectroscopy (1H-MRS) shows that high-altitude residents have altered whole brain pH and reduced inorganic phosphate to total phosphate (tP) ratios compared to persons dwelling at sea-level.28 In depressed patients, phosphorus MRS (31P-MRS) shows reduced nucleotide triphosphate (NTP) concentrations and decreased PCr concentrations; AD response is associated with increases in PCr and NTP.29 Hypoxia could also promote MDD by altering serotonin (5-HT) production. Chronic hypoxia reduces 5-HT in the forebrain and brainstem in rodents.30 The conversion of tryptophan to 5-hydroxytryptophan (5-HTP) by tryptophan hydroxylase is oxygen-dependent and slowed by hypoxia.31,32 Animal studies have shown that selective serotonin reuptake inhibitors (SSRIs) are not as effective at altitude,33 possibly because of inadequate 5-HT production. Reductions in 5-HT synthesis and inefficiencies in bioenergetics could both contribute to altered brain functional connectivity. MDD may disrupt cortical emotion regulation,34 and resting state functional connectivity (fcMRI) studies suggest that depression involves reduced connectivity between frontal cortical regions and the amygdala,35 while AD response correlates with normalization of those connections.36 Alterations in connectivity associated with AD response are correlated with changes in brain metabolites,37 suggesting a link to brain bioenergetics.

This suggests two natural supplements as interventions for depression. Oral creatine monohydrate (Cr) could improve bioenergetics in MDD, as Cr alters brain tCr, PCr, and NTP levels.38 Moreover, Cr produces improvements in mood39 correlated with normalization of PCr levels40 and structural connectivity.41 Alterations in 5-HT synthesis due to hypoxia could be rectified by 5-HTP, as its conversion to 5-HT is not oxygen-dependent. 5-HTP elevates brain 5-HT levels and has AD efficacy in clinical trials.42 The proposed study is a two-phase, three-armed trial to evaluate whether SSRI/SNRI augmentation with the supplements Cr, 5-HTP, or their combination (5-HTP+Cr) can enhance AD response in treatment-resistant MDD. In the R61 phase, the study will assess the ability of the interventions to alter biological signatures associated with depression, as measured by 31P-MRS, fcMRI, and changes in whole blood 5-HT. In the R33 phase, the study will attempt to replicate the above findings and evaluate their correlation with clinical outcomes. The study will have the following aims:

* Aim 1 (R61+R33): To identify 31P-MRS correlates of AD response in subjects with MDD receiving Cr, 5-HTP, or 5-HTP+Cr. It is hypothesized that subjects' frontal cortical metabolism will normalize compared to controls over 8 weeks in those receiving Cr or 5-HTP+Cr but not those receiving only 5-HTP.
* Aim 2 (R61+R33): To identify resting state fcMRI correlates of AD response in subjects with MDD receiving Cr, 5-HTP, or 5-HTP+Cr. It is hypothesized that resting functional connectivity in prefrontal regions will normalize (with improvement in hypoconnectivity between subgenual cingulate cortex and the remaining brain) over 8 weeks in all treatment groups compared to controls, with the greatest changes in the 5-HTP+Cr group.
* Aim 3 (R61+R33: To characterize changes in whole blood 5-HT levels in study participants. It is hypothesized that whole blood 5-HT will increase over 8 weeks in subjects receiving 5-HTP or 5-HTP+Cr, but not those receiving only Cr.
* Aim 4 (R33): To describe changes in HAM-D scores in study participants randomized between SSRI/SNRI augmentation with 5-HTP, Cr, or 5-HTP+Cr. It is hypothesized that HAM-D scores will improve over 8 weeks in all treatment groups, with the greatest changes in the 5-HTP+Cr group.

Study results will help elucidate the potential efficacy of a novel combination of nutritional supplements in persons with MDD, given strong epidemiologic and physiologic evidence suggesting that relative hypoxia can contribute to depression through alterations in brain bioenergetics and 5-HT synthesis. Target engagement will be indicated by improvements in functional connectivity and frontal cortical energy metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 25-40 years inclusive
* Current diagnosis of MDD identified by the SCID-5
* Current HAM-D17 score of > 16
* Adequate adherence to any FDA approved SSRI or SNRI for at least 8 weeks
* Right-handed
* Residing at > 4000 ft for at least 12 weeks

Exclusion Criteria:

* Any non-MDD and non-anxiety psychiatric diagnosis, as identified by the SCID-5
* History of or current diagnosis of renal disease, such as chronic renal failure, acute renal failure or end stage renal disease
* Current colitis or diverticulitis
* History of or current pulmonary disease
* Current smoking
* History of cardiac disease or QTc > 500ms
* History of fibromyalgia or any rheumatological condition
* History of or current seizure disorder
* Current serious suicide risk identified by the Columbia Severity Suicide Rating Scale
* Current treatment with an antipsychotic, mood stabilizer, or non-SSRI or SNRI antidepressant except for bupropion at FDA-approved doses or trazodone up to 200mg, or use of any supplements apart from standard multivitamins
* Positive pregnancy test, pregnancy, failure to use adequate birth control method
* Previous diagnosis of serotonin syndrome or evidence of serotonin syndrome
* Pre-existing eosinophilia (absolute eosinophil count > 500/uL)
* Contraindications to MRI: ferromagnetic implants, implanted devices, claustrophobia

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2024-03-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah Department of Psychiatry, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 5-HTP + Placebo | Creatine + Placebo | Creatine + 5-HTP | Double Placebo
Started | 11 | 10 | 11 | 11
Completed | 10 | 10 | 9 | 9
Not Completed | 1 | 0 | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 5-HTP + Placebo | Creatine + Placebo | Creatine + 5-HTP | Double Placebo | Total
Number analyzed (Participants) | 11 | 10 | 11 | 11 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.5 (5.5) | 35.5 (5.8) | 33.9 (4.9) | 30.8 (5.5) | 33.5 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 9 | 6 | 32
  Male | 3 | 1 | 2 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 10 | 9 | 11 | 10 | 40
  More than one race | 0 | 1 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: 17-Item Hamilton Depression Rating Scale Responders
Description: Hamilton Depression Rating Scale response rate: proportion of participants exhibiting >=50% reduction in baseline score; maximum possible score is 52, minimum possible score is 0. Higher scores suggest more severe depression.
Time Frame: 8 weeks
Population: The number of participants analyzed is less than the number of participants enrolled because of attrition in each group. Arm 1 lost one participant. Arm 2 lost one participant. Arm 3 lost two participants. Arm 4 lost two participants.
Measure: Count of Participants; unit: Participants
Arm/Group | 5-HTP + Placebo | Creatine + Placebo | Creatine + 5-HTP | Double Placebo
Number analyzed (Participants) | 10 | 9 | 9 | 9
Participants | 0 | 0 | 1 | 0

2. Secondary Outcome: Montgomery Asberg Depression Rating Scale Response Rate
Description: Montgomery Asberg Depression Rating Scale Response Rate. Proportion of responders. Response is a >=50% reduction in baseline score; minimum score 0; maximum score 60; higher scores suggest more severe depression
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 5-HTP + Placebo | Creatine + Placebo | Creatine + 5-HTP | Double Placebo
Number analyzed (Participants) | 10 | 9 | 9 | 9
Participants | 0 | 2 | 2 | 2

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | 5-HTP + Placebo | Creatine + Placebo | Creatine + 5-HTP | Double Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 5/11 | 3/10 | 4/11 | 4/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5-HTP + Placebo (N=11) | Creatine + Placebo (N=10) | Creatine + 5-HTP (N=11) | Double Placebo (N=11)
Nausea (Gastrointestinal disorders) | 4 (4) | 3 (3) | 4 (4) | 3 (3)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-07): https://cdn.clinicaltrials.gov/large-docs/83/NCT04395183/Prot_SAP_001.pdf